CLINICAL TRIAL: NCT01590771
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial in China to Study the Safety and Efficacy of the Addition of Sitagliptin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Sulfonylurea Therapy, Alone or in Combination With Metformin
Brief Title: A Study in China Evaluating the Safety and Efficacy of Adding Sitagliptin to Stable Therapy With Sulfonylurea With or Without Metformin in Participants With Type 2 Diabetes Mellitus (T2DM) (MK-0431-253)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0431-253
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Gliclazide; glimepiride; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin 100 mg once daily for 24 weeks. Participants will continue pre-study gliclazide or glimepiride with or without metformin for ≥10 weeks before and throughout the study. All participants will receive placebo during run-in period.
  Interventions: Drug: Sitagliptin; Drug: Gliclazide; Drug: Glimepiride; Drug: Metformin
- Placebo (Placebo Comparator): Matching placebo once daily for 24 weeks. Participants will continue pre-study gliclazide or glimepiride with or without metformin for ≥10 weeks before and throughout the study.
  Interventions: Drug: Placebo; Drug: Gliclazide; Drug: Glimepiride; Drug: Metformin

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg oral tablet once daily for 24 weeks
  Other Names: Januvia®; MK-0431
  Arms: Sitagliptin
Drug: Placebo — Matching placebo to sitagliptin oral tablet once daily for 24 weeks
  Arms: Placebo
Drug: Gliclazide — Participants will continue ongoing open-label therapy with gliclazide (dosed according to the China drug label) throughout the study.
Drug: Glimepiride — Participants will continue ongoing open-label therapy with glimepiride (dosed according to the China drug label) throughout the study.
Drug: Metformin — Participants will continue ongoing open-label therapy with metformin (at least 1500 mg daily) throughout the study.

SUMMARY:
A study to compare safety and efficacy of sitagliptin and placebo therapy when added to stable sulfonylurea alone or in combination with metformin in participants with type 2 diabetes mellitus (T2DM). The primary hypothesis of this study is that after 24 weeks, the addition of sitagliptin compared with placebo provides greater reduction in hemoglobin A1C (HbA1C) in T2DM participants on sulfonylurea alone or in combination with metformin.

ELIGIBILITY:
Inclusion Criteria:

* has T2DM
* is currently on a stable regimen of gliclazide or glimepiride, either alone or in combination with metformin for ≥ 10 weeks
* has a Visit 1/Screening HbA1C between 7.5% and 11.0%
* is a male, or a female who is highly unlikely to conceive during the study and for 14 days after the last dose of study medication

Exclusion Criteria:

* has a history of type 1 diabetes mellitus or a history of ketoacidosis
* has been treated with any antihyperglycemic therapies other than a sulfonylurea (alone or with metformin) within the prior 12 weeks or has ever

been treated with a dipeptidyl peptidase-4 inhibitor or a glucagon-like peptide-1 mimetic or analogue

* has a history of intolerance or hypersensitivity, or has any contraindication to sitagliptin, gliclazide/glimepiride, or metformin
* is on a weight loss program and not in the maintenance phase, or has started a weight loss medication or has undergone bariatric surgery within 12 months
* has undergone a surgical procedure within 4 weeks or has planned major surgery during the study
* has a medical history of active liver disease
* has had new or worsening signs or symptoms of coronary heart disease within the past 3 months, or has acute coronary syndrome, coronary artery intervention, or stroke or transient ischemic neurological disorder
* has a diagnosis of congestive heart failure with New York Heart Association Class III - IV cardiac status
* has a systolic blood pressure ≥ 160 mmHg or a diastolic blood pressure ≥ 90 mmHg
* has human immunodeficiency virus (HIV)
* has severe peripheral vascular disease
* is currently being treated for hyperthyroidism or is on thyroid hormone therapy and has not been on a stable dose for at least 6 weeks
* has a history of malignancy ≤ 5 years before the study, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* has a clinically important hematological disorder (such as aplastic anemia,

myeloproliferative or myelodysplastic syndromes, thrombocytopenia)

* is pregnant or breast feeding, or is expecting to conceive or donate eggs during the study, including 14 days after the last dose of study medication
* is a user of recreational or illicit drugs or has had a recent history of drug abuse

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2012-07-09 (Actual); Primary Completion 2014-06-10 (Actual); Study Completion 2014-06-24 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ba J, Han P, Yuan G, Mo Z, Pan C, Wu F, Xu L, Hanson ME, Engel SS, Shankar RR. Randomized trial assessing the safety and efficacy of sitagliptin in Chinese patients with type 2 diabetes mellitus inadequately controlled on sulfonylurea alone or combined with metformin. J Diabetes. 2017 Jul;9(7):667-676. doi: 10.1111/1753-0407.12456. Epub 2016 Sep 13. PMID 27502307
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0431-253&kw=0431-253&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants randomized population.
Groups:
- Sitagliptin: Sitagliptin 100 mg once daily for 24 weeks. Participants continued pre-study gliclazide or glimepiride with or without metformin for ≥10 weeks before and throughout the study.
- Placebo: Matching placebo once daily for 24 weeks. Participants continued pre-study gliclazide or glimepiride with or without metformin for ≥10 weeks before and throughout the study.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 249 | 249
Completed | 230 | 210
Not Completed | 19 | 39
Not completed — Other Protocol Specified Criteria | 5 | 14
Not completed — Withdrawal by Subject | 8 | 15
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 249 | 249 | 498
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (9.5) | 56.5 (9.3) | 57.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 117 | 249
  Male | 117 | 132 | 249
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent of glycosylated hemoglobin (A1C)] | 8.61 (1.06) | 8.48 (0.91) | 8.55 (0.99)
2-hour post meal glucose (2-hr PMG) [Mean (Standard Deviation); unit: mg/dL] — Sitagliptin, n=248; placebo, n=249; total, n=497
  mg/dL | 296.5 (68.0) | 290.2 (72.4) | 293.4 (70.2)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Sitagliptin, n=249; placebo, n=249; total, n=498
  mg/dL | 181.5 (40.9) | 179.8 (40.7) | 180.6 (40.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C Levels at Week 24 in Participants Receiving Sitagliptin and Sulfonylurea Alone or in Combination With Metformin
Description: A1C was measured as a percent. This change from baseline reflects the A1C percent at Week 24 minus the A1C percent at Week 0.
Time Frame: Baseline and Week 24
Population: Full analysis set consists of all participants who received at least one dose of study drug, have a baseline measurement, and have at least one post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of glycosylated hemoglobin (A1C)
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 243 | 236
Percent of glycosylated hemoglobin (A1C) | -0.88 [-0.99 to -0.76] | -0.27 [-0.38 to -0.15]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — The ANCOVA model controlled for treatment, metformin strata (on or not on metformin), and baseline A1C value; Robust regression = -0.61, 95% CI 2-sided [-0.77 to -0.44] — Based on robust regression using M-estimation with terms for treatment, metformin strata (on or not on metformin), and baseline A1C value

2. Secondary Outcome: Change From Baseline in 2-hr PMG Levels at Week 24 in Participants Receiving Sitagliptin and Sulfonylurea Alone or in Combination With Metformin
Description: This change from baseline reflects the 2-hr PMG level at Week 24 minus the 2-hr PMG level at Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 239 | 231
mg/dL | -40.7 [-49.4 to -31.9] | -7.7 [-16.6 to 1.2]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — The ANCOVA model controlled for treatment, metformin strata (on or not on metformin), and baseline 2-hr PMG value; Difference in least squares mean = -32.9, 95% CI 2-sided [-45.4 to -20.4]

3. Secondary Outcome: Change From Baseline in FPG Levels at Week 24 in Participants Receiving Sitagliptin and Sulfonylurea Alone or in Combination With Metformin
Description: This change from baseline reflects the FPG level at Week 24 minus the FPG level at Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 246 | 243
mg/dL | -24.4 (-29.1) [-29.1 to -19.8] | -7.7 [-12.3 to -3.0]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, Robust regression — Based on robust regression using M-estimation with terms for treatment, metformin strata (on or not on metformin), and baseline FPG value; Estimate difference = -16.8, 95% CI 2-sided [-23.3 to -10.2]

4. Secondary Outcome: Change From Baseline in A1C Levels at Week 24 in Participants Receiving Sitagliptin and Sulfonylurea in Combination With Metformin
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: Full analysis set (on metformin) consists of all participants on metformin who received at least one dose of study drug, have a baseline measurement, and have at least one post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of glycosylated hemoglobin (A1C)
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 111 | 112
Percent of glycosylated hemoglobin (A1C) | -0.86 [-1.01 to -0.71] | -0.45 [-0.60 to -0.30]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — The ANCOVA model controlled for treatment and baseline A1C value; Difference in least squares mean = -0.41, 95% CI 2-sided [-0.63 to -0.20]

5. Secondary Outcome: Change From Baseline in A1C Levels at Week 24 in Participants Receiving Sitagliptin and Sulfonylurea Alone
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: Full analysis set (not on metformin) consists of all participants not on metformin who received at least one dose of study drug, have a baseline measurement, and have at least one post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of glycosylated hemoglobin (A1C)
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 132 | 124
Percent of glycosylated hemoglobin (A1C) | -0.85 [-1.04 to -0.67] | -0.05 [-0.24 to 0.14]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — The ANCOVA model controlled for treatment and baseline A1C value; Difference in least squares mean = -0.80, 95% CI 2-sided [-1.07 to -0.53]

6. Secondary Outcome: Change From Baseline in 2-hr PMG Levels at Week 24 in Participants Receiving Sitagliptin and a Sulfonylurea in Combination With Metformin
Description: This change from baseline reflects the 2-hr PMG level at Week 24 minus the 2-hr PMG level at Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 109 | 111
mg/dL | -33.4 [-43.4 to -23.5] | -6.2 [-16.1 to 3.7]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, Robust regression — Based on robust regression using M-estimation with terms for treatment and baseline 2-hr PMG value; Estimate difference = -27.2, 95% CI 2-sided [-41.2 to -13.2]

7. Secondary Outcome: Change From Baseline in 2-hr PMG Levels at Week 24 in Participants Receiving Sitagliptin and Sulfonylurea Alone
Description: This change from baseline reflects the 2-hr PMG level at Week 24 minus the 2-hr PMG level at Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 130 | 120
mg/dL | -49.5 [-62.9 to -36.2] | -11.9 [-25.8 to 2.0]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — The ANCOVA model controlled for treatment and baseline 2-hr PMG value; Difference in least squares mean = -37.7, 95% CI 2-sided [-56.9 to -18.4]

8. Secondary Outcome: Change From Baseline in FPG Levels at Week 24 in Participants Receiving Sitagliptin and Sulfonylurea in Combination With Metformin
Description: This change from baseline reflects the FPG level at Week 24 minus the FPG level at Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 113 | 114
mg/dL | -22.2 [-28.4 to -16.0] | -5.7 [-11.9 to 0.5]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, Robust Regression — Based on robust regression using M-estimation with terms for treatment and baseline FPG value; Estimate Difference = -16.5, 95% CI 2-sided [-25.3 to -7.8]

9. Secondary Outcome: Change From Baseline in FPG Levels at Week 24 in Participants Receiving Sitagliptin and Sulfonylurea Alone
Description: This change from baseline reflects the FPG level at Week 24 minus the FPG level at Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 133 | 129
mg/dL | -26.3 [-33.3 to -19.4] | -9.3 [-16.3 to -2.3]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, Robust Regression — Based on robust regression using M-estimation with terms for treatment and baseline FPG value; Estimate Difference = -17.0, 95% CI 2-sided [-26.9 to -7.1]

10. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: An adverse event is any untoward medical occurrence in a participant administered study drug which does not necessarily have a causal relationship with the treatment. Adverse events may include the onset of new illness and the exacerbation of pre-existing conditions.
Time Frame: Up to 26 weeks
Population: All participants as treated population defined as all randomized participants who received at least one dose of study medication. Participants are included in the treatment group corresponding to the study treatment actually received.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 248 | 249
Participants | 106 | 98

11. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: as for outcome 10
Time Frame: Up to 24 weeks
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 248 | 249
Participants | 3 | 7

ADVERSE EVENTS:
Time Frame: Up to 26 weeks (including 14 days following the last dose of study medication).
Description: All participants as treated population defined as all randomized participants who received at least one dose of study medication. Participants are included in the treatment group corresponding to the study treatment actually received.
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 7/248 | 7/249
Other Adverse Events (participants affected / at risk) | 54/248 | 40/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=248) | Placebo (N=249)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=248) | Placebo (N=249)
Urinary tract infection (Infections and infestations) | 14 (14) | 11 (11)
Hyperlipidaemia (Metabolism and nutrition disorders) | 8 (8) | 15 (15)
Hypoglycaemia (Metabolism and nutrition disorders) | 35 (76) | 17 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding the study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.